CLINICAL TRIAL: NCT06774170
Title: Effect of Structured Follow-up Intervention on Glucose Status After Pancreatic Cancer Surgery: a Randomized Controlled Trial
Brief Title: Structured Follow-up Intervention on Glucose Status After Pancreatic Cancer Surgery
Acronym: FiGluR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Yaprak S. Ordin, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 223S838; TUBITAK (Other: The Scientific and Technological Research Council of Türkiye)
Record Dates: First submitted 2025-01-03; First posted 2025-01-14 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Pancreas Cancer; Diabetes
Keywords: pancreas cancer; pancreaticoduodenectomy; continuous glucose monitoring; type 3c diabetes mellitus; data mining
MeSH Terms: conditions — Pancreatic Neoplasms; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The study has a single-center, randomized, controlled, single-blind design. The study sample will include 40 patients (20 intervention group, 20 control group) with PD. The allocation ratio will be 1:1.
Who Masked: Participant
Masking Description: Participants do not know which group they are in. Both groups are included in the study in parallel. Both groups will be monitored continuously with a glucose device. The researcher will allocate equal time to both groups. Both groups will be called with the same frequency and the same time will be allocated for these interviews. The control group will receive routine post-operative training. The follow-up intervention initiative developed will be applied to the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Structured follow-up intervention will be performed
  Interventions: Behavioral: structured follow-up intervention
- Control group (No Intervention): Routine post-operative follow-up and education will be applied.

INTERVENTIONS:
Behavioral: structured follow-up intervention — The intervention has been created in light of the studies including type 1 and type 2 diabetes patients and experiences of the project team with patients after PD. Theoretical background of the intervention is based on the interventions developed for glucose management in type 1 and type 2 diabetes patients and the effect of the intervention will be evaluated by using the "plan-do-check-act" model.
  Arms: Intervention group

SUMMARY:
The primary aim of the present study is to examine the effect of a "structured follow-up intervention" to be performed in the first three months after PD on blood glucose. The exploratory aim of the study is to examine the effect of the "structured follow-up intervention" to be performed in the first three months after PD on patient outcomes (mortality, rehospitalization and having surgery, wound site complications, bile leakage, delayed gastric emptying, pancreatic fistula, myocardial infarct, cardiac arythmia, pneumonia, intraabdominal abscess, bleeding and pain) and the quality of life. The secondary aim of the study is to evaluate the factors affecting glucose levels in three months after PD by using data mining. Data mining will allow evaluation of all the factors affecting glucose levels by using detailed blood glucose predictors obtained through continuous glucose monitoring after PD. The study has a single-center, randomized, controlled, single-blind design. The study sample will include 40 patients with PD. The allocation ratio will be 1:1. Since being diagnosed as diabetes before surgery is an important variable, block randomization will be performed depending on whether the patients have the diagnosis of diabetes.

DETAILED DESCRIPTION:
The primary aim of the present study is to examine the effect of a "structured follow-up intervention" to be performed in the first three months after PD on blood glucose. The exploratory aim of the study is to examine the effect of the "structured follow-up intervention" to be performed in the first three months after PD on patient outcomes (mortality, rehospitalization and having surgery, wound site complications, bile leakage, delayed gastric emptying, pancreatic fistula, myocardial infarct, cardiac arythmia, pneumonia, intraabdominal abscess, bleeding and pain) and the quality of life. The secondary aim of the study is to evaluate the factors affecting glucose levels in three months after PD by using data mining. Data mining will allow evaluation of all the factors affecting glucose levels by using detailed blood glucose predictors obtained through continuous glucose monitoring after PD. The study has a single-center, randomized, controlled, single-blind design. The study sample will include 40 patients with PD. The allocation ratio will be 1:1. Since being diagnosed as diabetes before surgery is an important variable, block randomization will be performed depending on whether the patients have the diagnosis of diabetes.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for the particioants were; being over 18 years of age, being a smartphone user compatible with the Dexcom G6 application, having an internet connection, having a Mini Mental Test result of over 22 points for educated individuals and over 19 points for uneducated individuals, being willing to participate in the study, and having undergone pancreaticoduodenectomy.

In the study, "able to swallow table" is not eligibility criteria due to tablet (medication) adherence is not assssed In the study, patients with and without preoperative diabetes mellitus type II were included in the sample. Block randomization was performed according to the presence of DM. Therefore, the presence of diabetes is not an exclusion criterion.

In the literature, thyroid disease has not been identified as an exclusion criterion in studies related to pancreatogenic diabetes. The endocrinologist involved in this project did not find it necessary to add thyroid disease as an exclusion criterion.

Exclusion Criteria:

Exclusion criteria were; having developed sepsis after surgery, having been diagnosed with insulinoma, glycogonoma, ectopic ACTH syndrome before surgery, having been diagnosed with a psychiatric disease, clinical diagnosis of Alzheimer's Disease and being hospitalized.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Three months
  HbA1c
fasting blood glucose | Three months
  fasting blood glucose
mean glucose | Three months
  As a continuous glucose monitoring system, Decxom G6 will be utilized and blood glucose levels of the patients will be monitored for three months.
glucose standard deviation | Three months
  As a continuous glucose monitoring system, Decxom G6 will be utilized and blood glucose levels of the patients will be monitored for three months.
glucose variance coefficient | Three months
  As a continuous glucose monitoring system, Decxom G6 will be utilized and blood glucose levels of the patients will be monitored for three months.
GMI-glucose management indicator | Three months
  As a continuous glucose monitoring system, Decxom G6 will be utilized and blood glucose levels of the patients will be monitored for three months.
time spent at the target glucose value (Time in range) | Three months
  As a continuous glucose monitoring system, Decxom G6 will be utilized and blood glucose levels of the patients will be monitored for three months.

SECONDARY OUTCOMES:
rehospitalization/having surgery | Three months
  rehospitalization/having surgery
wound site complications | Three months
  wound site complications outcome will be collected from clinical data record
post-operative complications | Three months
  bile leakage, delayed gastric emptying, pancreatic fistula, myocardial infarct, cardiac arrythmia, pneumonia, intraabdominal abscess, bleeding outcomes as complications will be collected from clinical data record
pain | Three months
  Visual Analog Score for pain will be assessed. Pain will be assessed between 1-10 point; 1-no pian, 10-severe pain
quality of life-EORTC QOL-C30 | Three months
  Also quality of life of the patients will be assessed with European Organization for the Research and Treatment of Cancer Quality of life Questionnaire (EORTC QLQQ-C30) Version 3.0. All functional scales and individual item scores are transformed to a 0-100 scale with higher values indicating a higher functioning in functional scales and an increased presence of symptoms in symptom scales.
  Dear reviewer, there EORTC have 5 functional scales (physical functioning, role. functioning, emotional functioning, cognitive functioning, social functioning), global health status sub-scale, 9 symptom scales (fatigue, nause and vomiting, pain, dsypnoea, insomnia, apptite loss, constipation, diarhoea, financial difficulties). If we give each subscale, so much secondary outcomes and confused will be. Therefore we can not give each subscale as secondary outcomes.
quality of life-PAN26 | Three months
  Quality of life of pancreas cancer aspect will be assessed with PAN26. All functional scales and individual item scores are transformed to a 0-100 scale with higher values indicating a higher functioning in functional scales and an increased presence of symptoms in symptom scales.
  Dear reviewer, The QLQ-PAN26 consists of 15 sub-scales (pancreatic pain, bloating digestive symptoms, taste, indigestion, flatulence, weight loss, weakness arms and legs, dry mouth, hepatic symptoms, altered bowel habit, body image, taubled with side-effects, future worries and planning of activities) and 2 functional scales (satisfaction with health care, and sexuality). Because there are so many subsclaes, we prefer only PAN26 quality of lie aspect.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Balcova Inciralti, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No